CLINICAL TRIAL: NCT03776994
Title: A Phase 1 Dose Escalation Study to Assess the Safety and Immunogenicity of a Monovalent Virus-Like Particle (VLP) Venezuelan Equine Encephalitis Vaccine in Healthy Adults
Brief Title: Venezuelan Equine Encephalitis Monovalent Virus-Like Particle Vaccine
Acronym: VEEV
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: SRI International (Industry)
Collaborators: US Army Medical Research Institute of Infectious Diseases (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: SRI-VEEV-01
Record Dates: First submitted 2018-11-07; First posted 2018-12-17 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Encephalitis; Encephalitis, Viral; Infectious Encephalitis; Virus Diseases; Encephalomyelitis, Venezuelan Equine; Brain Diseases; Central Nervous System Diseases; Central Nervous System Viral Diseases; Alphavirus Infections; Togaviridae Infections; RNA Virus Infections; Central Nervous System Infections; Encephalomyelitis; Physiological Effects of Drugs; Vaccines; Encephalomyelitis, Equine; Nervous System Diseases
Keywords: Venezuelan Equine Encephalitis, vaccine; Intramuscular; Phase 1 clinical study
MeSH Terms: conditions — Encephalitis; Encephalitis, Viral; Infectious Encephalitis; Virus Diseases; Encephalomyelitis, Venezuelan Equine; Brain Diseases; Central Nervous System Diseases; Central Nervous System Viral Diseases; Alphavirus Infections; Togaviridae Infections; RNA Virus Infections; Central Nervous System Infections; Encephalomyelitis; Encephalomyelitis, Equine; Nervous System Diseases

STUDY DESIGN:
Intervention Model Description: To assess the safety and immunogenicity of a monovalent Venezuelan Equine Encephalitis (VEE) Virus-like Particle (VLP) Vaccine in healthy adults for protection against exposure to VEE virus (VEEV).
Who Masked: Participant
Masking Description: Subjects will be blinded to receiving the non-adjuvanted versus adjuvanted vaccines, but will not be blinded to the vaccine dosage. Vaccines will be brought into the subject rooms in a concealed container, and subjects will be asked to turn away from the dosing arm so that the SRI Clinical Trials' Unit (CTU) staff can prepare and administer the dose. Subjects may be unblinded if subject experiences a Serious Adverse Event (SAE) and upon notification to the data review team, called Protocol Safety Review Team (PSRT).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Group 1A 2 µg VEE Vaccine Alone (Experimental): Subgroup 1A, 2 µg VEE VLP Vaccine Alone Venezuelan equine encephalitis VLP Vaccine candidate
  Vaccinations on Day 0, Day 28, and Day 140
  Interventions: Biological: Vaccinations on Day 0, Day 28, and Day 140
- Group 2A 10 µg VEE Vaccine Alone (Experimental): Venezuelan equine encephalitis VLP Vaccine candidate Subgroup 2A, 10 µg VLP Vaccine Alone
  Vaccinations on Day 0, Day 28, and Day 140
  Interventions: Biological: Vaccinations on Day 0, Day 28, and Day 140
- Group 3A 20 µg VEE Vaccine Alone (Experimental): Venezuelan equine encephalitis VLP Vaccine candidate Subgroup 3A, 20 µg VEE VLP Vaccine Alone
  Vaccinations on Day 0, Day 28, and Day 140
  Interventions: Biological: Vaccinations on Day 0, Day 28, and Day 140
- Group 1B 2 µg VEE Vaccine and Adjuvant (Experimental): Venezuelan equine encephalitis VLP Vaccine candidate with Adjuvant Subgroup 1B, 2 µg VEE VLP Vaccine with Adjuvant (Adjuvant - Aluminum hydroxide, 5 mg/mL)
  Vaccinations on Day 0, Day 28, and Day 140
  Interventions: Biological: Vaccinations on Day 0, Day 28, and Day 140
- Group 2B 10 µg VEE Vaccine with Adjuvant (Experimental): Venezuelan equine encephalitis VLP Vaccine candidate with Adjuvant Subgroup 2B, 10 µg VEE VLP Vaccine with Adjuvant (Adjuvant - Aluminum hydroxide, 5 mg/mL)
  Vaccinations on Day 0, Day 28, and Day 140
  Interventions: Biological: Vaccinations on Day 0, Day 28, and Day 140
- Group 3B 20 µg VEE Vaccine with Adjuvant (Experimental): Venezuelan equine encephalitis VLP Vaccine candidate with Adjuvant Subgroup 3B, 20 µg VEE VLP Vaccine with Adjuvant (Adjuvant - Aluminum hydroxide, 5 mg/mL)
  Vaccinations on Day 0, Day 28, and Day 140
  Interventions: Biological: Vaccinations on Day 0, Day 28, and Day 140

INTERVENTIONS:
Biological: Vaccinations on Day 0, Day 28, and Day 140 — The monovalent VEE VLP vaccine (the same VEE VLP study agent which comprises the VEE portion of the NIAID trivalent alphaviral VLP vaccine) will use the same vaccination regimen (Day 0, Week 4 [Day 28], and Week 20 [Day 140]) and the vaccine dosages (2 μg, 10 μg, and 20 μg)

SUMMARY:
The primary objective of the study is to evaluate the safety and immunogenicity of non-adjuvanted and adjuvanted monovalent VEE VLP Vaccine in healthy adults (ages 18-50 years) when administered via intramuscular (IM) injection at escalating doses of 2 μg, 10 μg, and 20 μg as a 2-dose primary series (Day 0, Day 28) with a Day 140 booster dose. The secondary objective of the study is to evaluate immunogenicity of the vaccine at the aforementioned time points

DETAILED DESCRIPTION:
This Phase 1 dose escalation study will evaluate safety and immunogenicity of both non-adjuvanted and adjuvanted VEE VLP vaccine in three dose groups (2 μg, 10 μg, and 20 μg) given as a 2-dose primary series IM injection (Days 0 and Week 4 [Day 28]) followed by a booster dose injection (Week 20 [Day 140]). Each group will consist of 30 subjects, for a total of 90 study subjects. Each group of 30 subjects will be randomized to receive either non-adjuvanted vaccine (Subgroup A; n=15) or adjuvanted vaccine (Subgroup B; n=15). Subjects will be blinded to receiving the non-adjuvanted versus adjuvanted vaccine, but will not be blinded to the vaccine dosage. Enrollment will utilize a sentinel dose design, with only one subject receiving a vaccine dose the initial day, 2 subjects the following day, and 3 subjects the subsequent day, before proceeding with further enrollments in that group. Subjects in each Group will be randomized to receive the vaccine dose either without adjuvant (Subgroup A) or with adjuvant (Subgroup B).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between the ages of 18 and 50.
2. Understanding of the requirements of the study, provision of written informed consent, and agreement to abide by the study restrictions.
3. In good general health (no chronic health condition) and an acceptable medical history, physical examination and screening laboratory studies within 28 days of enrollment on the study (specific laboratory requirements are listed below).
4. Negative urine screen for drugs of abuse at screening.
5. Body weight ≥ 49.8 kg and ≤ 110 kg. If body weight is over 110 kg, then body mass index (BMI) will be considered and must be < 40 kg/m2. The National Institutes of Health National Heart, Lung, and Blood Institute BMI calculator will be used to make this determination (https://www.nhlbi.nih.gov/health/educational/lose_wt/BMI/bmi-m.htm).
6. Available for entire clinical study duration of 44 weeks.
7. Individual agrees to not receive non-study vaccines during study unless urgent medical indication (i.e., tetanus booster, rabies vaccine).
8. Females must be of non-childbearing potential or agree to use two types of an acceptable form of FDA-approved contraception through the duration of the study and must not be pregnant or lactating. If volunteers are sexually abstinent, they are not required to use additional forms of birth control. Non-childbearing potential is defined as being post-menopausal (absence of menses for 12 consecutive months not caused by drugs or hormones), status after bilateral tubal ligation for at least 1 year, status after bilateral oophorectomy, or status after hysterectomy. Examples of acceptable forms of birth control include but are not limited to barrier methods, Depo-Provera®, Norplant®, Nova Ring®, Ortho Evra® (birth control patch), and oral contraceptives. Absence of pregnancy in women of child-bearing potential (WOCBP) is indicated by a negative history of current pregnancy, a negative urine pregnancy test at screening, and a negative urine pregnancy test performed within 1 day before each administration of study vaccine.

Exclusion Criteria:

Laboratory Studies:

Any clinically significant hematology, chemistry, coagulation, serology, or urinalysis value on screening labs (some examples are listed below):

* Hemoglobin <11.5 g/dL for women; <12.0 g/dL for men
* White blood cell (WBC) Count <3,000 or >13,000/mm3
* Total lymphocyte count <800 cell/ mm3
* Platelets <125,000 or >500,000/mm3
* Alanine aminotransferase (ALT) >1.2 upper limits of normal
* Serum creatinine not greater than the upper limits of normal
* Prothrombin Time (PT) >12.5 seconds
* International Normalized Ratio (INR) >1.32
* Partial Thromboplastin Time (PTT) >36.5 seconds
* Positive urine pregnancy test
* HBsAg positive, or serologic evidence of infection with Hepatitis C (HCV) or Human Immunodeficiency Virus (HIV)

Subject has a history of any of the following:

1. Active substance or alcohol abuse (within the previous 2 years as per the judgment of the investigator).
2. History of any psychiatric condition (e.g., past or present psychoses) that could jeopardize the subject's safety or the subject's ability to comply with the protocol.
3. History of a significant medical condition that could jeopardize the subject's safety or the subject's ability to comply with the protocol. Exclusionary medical conditions include (but not limited to) significant endocrine disorders (e.g., diabetes mellitus, type I or II), gastrointestinal disorders (e.g., active peptic ulcer disease, hepatitis), hematological disease (e.g., thrombocytopenia, diathesis, coagulopathy, asplenia or functional asplenia), renal disease (e.g., acute or chronic), neurological disease (e.g., seizure disorder other than a history of febrile seizures, or seizures secondary to alcohol withdrawal >3years ago, or seizures that have not required treatment within the last 3 years, history of Guillain-Barré syndrome), pulmonary disease (e.g., including asthma or chronic obstructive pulmonary disease (COPD) that is unstable or required emergent care, urgent care, hospitalization or intubation during the past two years and that is expected to require the use of oral or intravenous corticosteroids), autoimmune disorders, active malignancy (or previous malignancy and at risk for disease recurrence or malignancy for which there is no reasonable assurance of sustained cure, or likely to recur during the period of the study), cardiac disorders (e.g., congestive heart failure), and other significant conditions as deemed by the investigator to be an exclusion from the study.
4. Recipient of an organ transplant (solid or hematopoietic)

Subject has received any of the following substances:

1. Administration of blood products within 16 weeks and immunoglobulin products within 8 weeks preceding enrollment or planned vaccine administration during the study period.
2. Prior alphaviral vaccines (VEE, Eastern equine encephalitis (EEE), western equine encephalitis (WEE), or chikungunya) or VEE subunit vaccinations.
3. Investigational vaccine in the previous 6 months before receiving the initial vaccine dose of this study (or plans to receive during the study).
4. Marketed medically indicated subunit or inactivated vaccines (i.e., influenza, pneumococcal vaccines) or allergy antigen injections) within 28 days after or within 28 days before any study vaccine doses.
5. Marketed attenuated vaccines (i.e., measles, rubella) within 28 days after or within 28 days before any study vaccine doses.
6. Investigational drug within 30 days of enrollment.
7. Current tuberculosis prophylaxis or therapy or current HIV prophylaxis.
8. Systemic immunosuppressive or cytotoxic medications within 12 weeks prior to enrollment [does not exclude individuals who received a short course of corticosteroids (<10 days duration or a single injection) for a self-limited condition greater than at least 2 weeks prior to enrollment].

Subject has a history of the following:

1. History of a serious reaction to vaccines that preclude receipt of study vaccine as determined by the investigator
2. Allergy to vaccine, vaccine components or aluminum compounds.
3. History of serious allergic reactions or anaphylaxis (e.g., vaccines, insect stings, food, drugs, or other biological products).
4. Febrile illness or significant infection at the time of vaccination (may be rescheduled for enrollment). Must be afebrile for 72 hours prior to receiving vaccine as reported by the subject to the SRI Clinical Trials' Unit (CTU) staff.
5. A confirmed or suspected history of VEEV or other alphaviral infection (i.e., eastern equine encephalitis (EEE), western equine encephalitis (WEE), chikungunya) or other encephalitis infection or a history of employment in a laboratory that worked with VEE virus (VEEV).
6. Bleeding disorder (e.g., factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or history of significant bruising or bleeding difficulties with IM injections or blood draws.
7. Blood donation within 60 days of enrollment. -

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2018-07-17 (Actual); Primary Completion 2020-07-27 (Actual); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Number of subjects reporting solicited local adverse events | Through the study duration of 44 weeks
  • The solicited local adverse events (SLAEs) are specified and collected in daily diary questionnaires for 1 week after each vaccination in each arm of the study (Days 0-7, 28-35, and 140-147). These SLAEs include pain, tenderness, induration or swelling, and erythema. Symptoms are counted once if subjects experienced the symptom at any severity during the reporting period. The number of local symptoms is the total of one or more local symptom at any severity. The severity of the SLAEs will be graded as Mild (Grade 1), Moderate (Grade 2), Severe (Grade 3) or Potentially Life Threatening (Grade 4). SLAEs will be characterized according to the "Toxicity grading scale for healthy adult and adolescent volunteers enrolled in preventative vaccine trials" FDA Guidance for Industry (Sept 2007). The frequency of SLAEs will each be expressed as the number of subjects experiencing these adverse events for the 3 vaccinations within each of the 6 arms of the study.
Number of subjects reporting solicited systemic adverse events | Through the study duration of 44 weeks
  • The solicited systemic adverse events (SSAEs) are specified and collected in daily diary questionnaires for 1 week after each vaccination in each arm of the study (Days 0-7, 28-35, and 140-147). These SSAEs are fever, malaise, myalgia, arthralgia, headache, chills, fever, nausea, and rash. Symptoms are counted once if subjects experienced the symptom at any severity during the reporting period. The number of systemic symptoms is the total of one or more systemic symptom at any severity. The severity of the SSAEs will be graded as Mild (Grade 1), Moderate (Grade 2), Severe (Grade 3) or Potentially Life Threatening (Grade 4). SSAEs will be characterized according to the "Toxicity grading scale for healthy adult and adolescent volunteers enrolled in preventative vaccine trials" FDA Guidance for Industry (Sept 2007). The frequency of SSAEs will each be expressed as the number of subjects experiencing these adverse events for the 3 vaccinations within each of the 6 arms of the study.
Number of subjects reporting treatment-emergent adverse events | Through the study duration of 44 weeks
  • Unsolicited treatment-emergent adverse events (collected for 28 days after each vaccination or Days 0-28, Days 28-56, and Days 140-168) will be collected and tabulated. MedDRA version 21.0 will be used for coding. The number of subjects experiencing the unsolicited treatment-emergent adverse events within the 28 days after the three vaccinations will be reported for each of the six arms.
Number of subjects reporting serious adverse events | Through the study duration of 44 weeks
  • Serious adverse events will be collected throughout the study. The frequency of these solicited adverse events will each be expressed as the number of subjects experiencing these adverse events for the three vaccinations within each of the six arms of the study.
Number of subjects with abnormalities in serum creatinine concentrations | Through the study duration of 44 weeks
  • Serum creatinine is measured on Days 0, 7, 28, 35, 56, 140, 147, 168 and 308. The normal range for adults aged 18-50 years for men is 0.6 - 1.35 mg/dL and women 0.50 - 1.10 mg/dL. The abnormal serum creatinine values are characterized as follows: Grade 1 (1.5 - 1.7 mg/dL), Grade 2 (1.8 - 2.0 mg/dL), Grade 3 (2.1 - 2.5 mg/dL), and grade 4 (>2.5 mg/dL or requires dialysis) according to the "Toxicity grading scale for healthy adult and adolescent volunteers enrolled in preventative vaccine trials" FDA Guidance for Industry (September 2007). The frequency and severity of these adverse events will be expressed as the number of subjects with any abnormal result for the three vaccinations within each of the six arms of the study.
Number of subjects with abnormal serum alanine aminotransferase concentrations | Through the study duration of 44 weeks
  • Serum alanine aminotransferase is measured on Days 0, 7, 28, 35, 56, 140, 147, 168 and 308.The normal range for adults ages 18-50 years for men is 9 - 46 mg/dL and women 6 - 29 mg/dL. The grading is characterized as follows: Grade 1 (1.1 - 2.5 x upper limits of normal [ULN]), Grade 2 (2.6 - 5.0 ULN), Grade 3 (5.1 - 10 x ULN) and Grade 4 (>10 x ULN) according to the "Toxicity grading scale for healthy adult and adolescent volunteers enrolled in preventative vaccine trials" FDA Guidance for Industry (September 2007). The frequency and severity of these adverse events will be expressed as the number of subjects with any abnormal result for the three vaccinations within each of the six arms of the study.
Number of subjects with abnormal complete blood counts | Through the study duration of 44 weeks
  • Complete blood count is measured on Days 0, 7, 28, 35, 56, 140, 147, 168 and 308. The changes (either increases or decreases) in components of the complete blood count (e.g., hemoglobin, hematocrit, total white blood cell to and differential, and platelet count) are tabulated according to Grades 1- 4 in the "Toxicity grading scale for healthy adult and adolescent volunteers enrolled in preventative vaccine trials" FDA Guidance for Industry (September 2007). The frequency and severity of any abnormal results will be expressed as the number of subjects with any abnormal result for the three vaccinations within each of the six arms of the study.

SECONDARY OUTCOMES:
Number of subjects with neutralizing antibody titers as assessed by a plaque reduction neutralization test (PRNT50) | Through the study duration of 44 weeks
  • The number of subjects with detectable titers of neutralization antibodies will be measured with the plaque reduction neutralization test (PRNT50) at four weeks after the second injection (Week 8), four weeks after the third injection (Week 24) and at the end of the study (Week 44). The titers of the anti-VEEV neutralizing antibodies will be expressed as a geometric mean titer for the three vaccinations within each of the six arms of the study
The duration of detectable neutralizing antibody titers as assessed by the plaque reduction neutralization test (PRNT50) | Through the study duration of 44 weeks
  • The duration of detectable titers of neutralization antibodies in subjects will be measured with the plaque reduction neutralization test (PRNT50) at four weeks after the second injection (Week 8), four weeks after the third injection (Week 24) and at the end of the study (Week 44, Day 308). The titers of the anti-VEEV neutralizing antibodies will be expressed as a geometric mean titer for the three vaccinations within each of the six arms of the study
The magnitude of neutralizing antibodies as assessed by a plaque reduction neutralization test (PRNT50) | Through the study duration of 44 weeks
  • The magnitude of detectable titers of neutralization antibodies in subjects will be measured with the plaque reduction neutralization test (PRNT50) at four weeks after the second injection (Week 8), four weeks after the third injection (Week 24) and at the end of the study (Week 44, Day 308). The titers of the anti-VEEV neutralizing antibodies will be expressed as a geometric mean titer for the three vaccinations within each of the six arms of the study

CONTACTS AND LOCATIONS:
Overall Officials: Sascha Goonewardena, MD, Principal Investigator — SRI International
Locations (1):
- SRI Biosciences Clinical Trials Unit, Plymouth, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hoke CH Jr. History of U.S. military contributions to the study of viral encephalitis. Mil Med. 2005 Apr;170(4 Suppl):92-105. doi: 10.7205/milmed.170.4s.92. PMID 15916288
- [Background] Tyler KL. Acute Viral Encephalitis. N Engl J Med. 2018 Aug 9;379(6):557-566. doi: 10.1056/NEJMra1708714. No abstract available. PMID 30089069
- [Background] Paessler S, Weaver SC. Vaccines for Venezuelan equine encephalitis. Vaccine. 2009 Nov 5;27 Suppl 4:D80-5. doi: 10.1016/j.vaccine.2009.07.095. PMID 19837294